CLINICAL TRIAL: NCT06248099
Title: A Bioequivalence Study of Nebivolol Tablets 5 mg Relative to Nebilet Tablets 5 mg in Healthy Thai Volunteers Under Fasting Condition
Brief Title: Nebivolol Tablets 5 mg Relative to Nebilet Tablets 5 mg
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bio-innova Co., Ltd (Industry)
Responsible Party: Principal Investigator, Sasitorn Kittivoravitkul, Principal Investigator, Bio-innova Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NEB-027-23
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Healthy Subjects
Keywords: Bioequivalence Nebivolol tablets 5 mg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1-Nebivolol test product and then reference product (Experimental): Participants will receive treatment 1 in period 1 and treatment 2 in period 2. Where treatment 1= Nebivolol tablets 5 mg test product, treatment 2= Nebivolol tablets 5 mg reference product.
  Interventions: Drug: Nebivolol-Test product
- Sequence 2-Nebivolol reference product and then test product (Experimental): Participants will receive treatment 2 in period 1 and treatment 1 in period 2. Where treatment 1= Nebivolol tablets 5 mg test product, treatment 2= Nebivolol tablets 5 mg reference product.
  Interventions: Drug: Nebivolol-Reference product

INTERVENTIONS:
Drug: Nebivolol-Test product — Test-Product: Nebivolol tablets 5 mg Manufactured by: Hetero Labs Limited, India
  Arms: Sequence 1-Nebivolol test product and then reference product
Drug: Nebivolol-Reference product — Reference-product: Nebilet tablets 5 mg Manufactured by: BERLIN CHEMIE AG, Germany
  Arms: Sequence 2-Nebivolol reference product and then test product

SUMMARY:
The study is to compare the rate and extent of absorption of a generic formulation with that of a reference for mulation when given as equal labeled dose. The study will be randomized, open-label, single dose, two way crossover design with two-period, two-treatment and two-sequence under fasting condition and at least 28 days washout period between the doses.

DETAILED DESCRIPTION:
Title A Bioequivalence study of a randomized, open-label, single dose, two-way crossover design with two-period, two-treatment, and two-sequence of Nebivolol tablets 5 mg relative to Nebilet tablets 5 mg in healthy Thai volunteers under fasting condition

Objectives The primary objective is to compare the rate and extent of absorption of a generic formulation with that of a reference formulation when given as equal labeled dose. The secondary objective is to evaluate the safety after oral administration of both test and reference formulation in healthy Thai volunteers.

Study Design Randomized, open-label, single dose, two-way crossover design with two-period, two-treatment, and two-sequence under fasting condition

Sample Size 46 Healthy Human Thai subjects. Four extra subjects if available, may be checked-in on the day of check in of period-I to compensate for any dropout prior to dosing of period-I. These subjects will be dosed if there are dropouts prior to dosing in period-I. If there are no dropouts, these subjects will be checked-out without being dosed after completion of dosing in period-I.

Drug-Product Test-Product: Nebivolol tablets 5 mg

Reference-product: Nebilet tablets 5 mg Manufactured by: BERLIN CHEMIE AG, Germany

Administration After an overnight fasting at clinical facility of at least 10 hours, each volunteer will receive a single dose of Nebivolol tablets 5 mg of either test or reference with 250 mL of drinking water. Each volunteer will be allowed to drink water as desire except 1 hour before and after drug administration. The formulation is given in a crossover fashion as per the randomization schedule. After the administration, the subject's oral cavity will be checked by using flashlight to confirm complete medication and fluid consumption by pharmacist.

Blood Schedule In each period, a total of 24 blood samples (approximately 7 mL each) will be collected pre-dose (0.000 hour) and at 0.167, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.500, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000, 60.000 and 72.000 hours after study drug administration, respectively. The sample collection at 36.000, 48.000, 60.000 and 72.000 hours after dosing will be on ambulatory basis (i.e. on separate visit).

Sample Collection Blood samples will be collected through an indwelling catheter placed in a vein using disposable syringe or through fresh venipuncture with disposable syringes and needles. Approximately 7 mL blood sample will be withdrawn and transferred to sample collection pre-labeled tubes containing K3EDTA as anticoagulant at each sampling time point. After collection of blood samples from each subject at each time point, samples will be centrifuged at 4000 rpm for 5 minutes at 4±2°C. After centrifugation, the plasma samples will be aliquot into two pre-labeled cryovials for approximately 1 mL per each cryovial. Cryovials containing plasma sample will be stored at -70±10 °C.

Analytical Method Nebivolol plasma concentration will be assayed as per international Guidelines/In-house SOP by using a UPLC-MS/MS method.

Pharmacokinetic Parameters Primary pharmacokinetic parameter: Cmax, AUC0→t and AUC0→∞ and secondary pharmacokinetic parameter: Tmax, T1/2, Kel, AUC0→t/AUC0→∞ will be determined from the plasma concentration data of analytes.

Statistical Analysis ANOVA, two one-sided tests for bioequivalence, for log-transformed pharmacokinetic parameters Cmax, AUC0→t and AUC0→∞ will be performed.

Acceptance Criteria for Bioequivalence To be considered as bioequivalent, the 90% Confidence Interval of the geometric means ratio of Cmax, AUC0→t and AUC0→∞ of Nebivolol of test and reference products should be in the interval of 80.00-125.00% for the log-transformed data.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent prior to participate in the study.
2. Healthy Thai subjects are between 18 to 55 years of age.
3. The Body Mass Index (BMI) ranges from 18.5 to 30 kg/m2.
4. Comprehensive of the nature and purpose of the study and compliance with the requirement of the entire protocol and allow investigators to draw 7 mL of blood for monitoring subjects' safety after the completion of the study.
5. Negative urine pregnancy test for women and no breast-feeding.
6. Absence of significant diseases or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or surgery during the screening. Some of the laboratory values e.g. Complete blood count etc. that out of the normal range will be carefully considered by physician.

Exclusion Criteria:

1. History or evidence of allergy or hypersensitivity to Nebivolol or Beta-blockers or any of the excipients of this product.
2. Subject with B.P. is Systolic B.P < 100, ≥ 140 mm/Hg, Diastolic B.P < 70, ≥ 90 mm/Hg or pulse rate > 100 beats per minute.
3. Serum bilirubin greater than 1.5 times the upper limit of reference range (ULRR).*
4. Serum creatinine greater than 1.5 times the upper limit of reference range (ULRR).*
5. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2 times the upper limit of reference range (ULRR).*
6. Positive of hepatitis B or C virus.
7. Have more than one abnormal EKG, which is considered as clinically significant. *
8. History of hyperthyroidism
9. History or evidence of heart, renal, hepatic disease, pulmonary obstructive disease, bronchial asthma, hypertension or glaucoma
10. History or evidence of gastrointestinal disorder likely to influence drug absorption or previous GI surgery other than appendectomy.
11. Any major illness in the past 3 months or any significant ongoing chronic medical illness.
12. History of psychiatric disorder.
13. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for males (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) and cannot stop at least 2 days before the study drug administration and until the completion of each period of the study.
14. History of usually smoking (more than 10 cigarettes per day within past 1 year), if moderate smokers (less than 10 cigarettes per day) cannot stop at least 7 days before the study drug administration and until the completion of each period of the study.
15. High caffeine consumption (more than 5 cups of coffee or tea per day) and cannot stop at least 2 days before the study drug administration and until the completion of each period of the study.
16. Positive drug abused test in urine (Benzodiazepines, Marijuana (THC), Methamphetamine, Cocaine and Opioids).
17. Receipt of any prescription drug therapy within 14 days or 5 half-lives (whichever longer) preceding the first dose of study medication or over-the-counter (OTC) drugs or herbal medicines/food supplement within 7 days or hormonal methods of contraception within 28 days (Depo-Provera must be discontinued at least 6 months) prior to receiving the first dose of study medication.
18. History of difficulty in accessibility of veins in left and right arm.
19. Blood donation (one unit or 450 mL) within the past 3 months before the study.
20. Participation in any clinical study within the past 3 months before the study.
21. Subjects who are unwilling or unable to comply with the lifestyle guidelines described in this protocol.

(* Depend on decision of principal investigator and/or clinical investigator)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-07-09 (Estimated); Primary Completion 2024-08-17 (Estimated); Study Completion 2024-09-14 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC 0-t) | Blood samples will be collected for PK analyses in each period pre-dose and at 0.167, 0.333, 0.50, 0.750, 1.00, 1.250, 1.50, 1.750, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 36.00, 48.00, 60.00 and 72.00 hour post-dose
  pre-dose (0.00 hour) and at 0.167, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.500, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000, 60.000 and 72.000 hours post-dose
Maximal measured plasma concentration (Cmax) | Blood samples will be collected for PK analyses in each period pre-dose and at 0.167, 0.333, 0.50, 0.750, 1.00, 1.250, 1.50, 1.750, 2.00, 2.50, 3.00, 3.50, 4.00, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 36.00, 48.00, 60.00 and 72.00 hour post-dose
  pre-dose (0.00 hour) and at 0.167, 0.333, 0.500, 0.750, 1.000, 1.250, 1.500, 1.750, 2.000, 2.500, 3.000, 3.500, 4.000, 5.000, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000, 60.000 and 72.000 hours post-dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | Approximately the day 28 after the last visit
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

IPD SHARING:
Plan to Share IPD: No
Company Policy